CLINICAL TRIAL: NCT01440751
Title: Comparative Study of the Safety and Effectiveness of Ologen Collagen Matrix Versus Mitomycin-C in Glaucoma Filtering Surgery
Brief Title: Comparative Study of Ologen Collagen Matrix Versus Mitomycin-C in Glaucoma Filtering Surgery
Acronym: MCToCM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aeon Astron Europe B.V. (Industry)
Collaborators: The New York Eye & Ear Infirmary (Other); Robert Ritch, MD, LLC. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAE-CT-USA-2010-02
Record Dates: First submitted 2011-09-14; First posted 2011-09-27 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma
Keywords: ologen collagen matrix; mitomycin-C; trabeculectomy; glaucoma; filtering surgery
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ologen Collagen Matrix (Experimental): When performing glaucoma surgery, a trabeculectomy, use ologen Collagen Matrix instead of MMC before closing the conjunctiva
  Interventions: Device: Use of ologen Collagen Matrix in trabeculectomy (ologen)
- Mitomycin-C (MMC) (Active Comparator): When performing glaucoma surgery, a trabeculectomy, use MMC as antifibrotic agent before closing the conjunctiva
  Interventions: Drug: Use of Mitomycin-C (MMC) in trabeculectomy

INTERVENTIONS:
Device: Use of ologen Collagen Matrix in trabeculectomy (ologen) — Place ologen CM on the top of the loosely-sutured scleral flap under conjunctiva before suturing. It is recommended to suture the scleral flap with 1 or 2 stiches loosely for the convenience of future suture lysis and to coordinate with the tamponading effect of ologen CM to create a fluctuating scleral flap that prevents bleb wound adhesion and modulates aqueous humor outflow for ideal IOP control without leakage.
  Arms: ologen Collagen Matrix
Drug: Use of Mitomycin-C (MMC) in trabeculectomy — After outlining and creating a superficial scleral flap, a cellulose sponge soaked with MMC(0.4mg/mL) is applied for up to 3 mins according to physician's routine method of application. The area treated is copiously irrigated with balanced isotonic solution. Alternatively, 15mcg of MMC may be injected intra-Tenon's at the end of the procedure. Patients receiving mitomycin will be billed as per operating room practice.
  Arms: Mitomycin-C (MMC)

SUMMARY:
The objective of this prospective randomised study is to compare the efficacy and safety of ologen CM (Collagen matrix) and Mitomycin-C (MMC) as adjuncts to filtration surgery in uncontrolled treated glaucoma cases, the efficacy being the primary objective and the safety being the secondary.

DETAILED DESCRIPTION:
"ologen ® CM" is a biodegradable collagen matrix. To prevent episcleral fibrosis and subconjunctival scarring thay may result in the surgical failure in trabeculectomy, its sporous matrix modulates the migrations and proliferations of fibroblasts to create a vascular and long-lasting bleb without the adverse effects, such as avascular thin bleb wall, bleb leak, hypotony, and inflammations, potentially caused by the regeneration suppression effects upon the use of cytotoxic agents as anti-fibrotic agents, such as MMC (Mitomycin-C)in the study.

Results of ologen CM studies have been published at conferences and published in peer-reviewed journals; ologen CM is approved in Europe as an aid for tissue repair, and by the FDA in the US as an adjunct in wound management(K080868). In general, over 6,000 ologen CM have been implanted worldwide during the past two years with good results and excellent safety profile.

The clinical trial is a phase-IV post-marketing FDA approved device study designed as open-label, randomised, parallel, and comparative. 128 patients at 8 sites are anticipated to be recruited according to the enrollment criteria, while randomisation will be assigned by a sealed envelope system after the patient has signed consent. Trabeculectomy is performed thereafter with either MMC or ologen CM applications as described in the protocol with postoperative parameters to be measured and analysed with non-parametric tests(Chi-square, Fisher's exact, Wilcoxon, and Mann-Whitney tests) as well as Kaplan-Meier survival models.

ELIGIBILITY:
Inclusion Criteria:

* Age > 30 years (inclusive)
* Uncontrolled treated glaucoma requiring trabeculectomy
* Subject must be able and willing to cooperate with investigation plan
* Subject must be able and willing to complete postoperative follow-up requirements
* subject must be willing to sign informed consent form

Exclusion Criteria:

* Known allergic reaction to MMC or porcine collagen
* Neovascular, uveitic, aphakic glaucoma, previous incisional glaucoma surgery
* Prior cataract unless clear corneal incision
* Previous conjunctival or strabismus surgery
* Participation in an investigational study during 30 days prior to trabeculectomy
* Ocular infection within 14 days prior to trabeculectomy
* Pregnant or breast-feeding women

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure(IOP) reduction | At postoperative up to 24 months.
  "Complete success" is consider for IOP less than 21mmHg(inclusive) with no glaucoma medications and with more than 20% reduction(inclusive) from baseline IOP.
  Definition of success rate is calculated in percentage by the number of complete success patients over the total sample size.
  "Qualified success" that meets the postoperative IOP requirements with postoperative glaucoma medicaitons and "Failure" of meeting the IOP requirements are the other efficacy parameters.
  In the specified time frame, patients will also visit for record at day 1, 7, 14, 30, 90, 180 days, 12, 18, and 24 months.

SECONDARY OUTCOMES:
Postoperative complications and appearances | At postoperative up to 24 months.
  Inspections of hyphema, severe anterior chamber reaction, hypotony, supercholoidal hemorrhage, flat anterior chamber, endophthalmitis, choroidal detachment, wound or bleb leak.
  Visual acuity, bleb appearance, and anterior chamber inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — Robert Ritch, MD, LLC.; Steven Sarkisian, MD, Study Director — Dean McGee Eye Institute; Robert Fechtner, MD, Study Director — Institute of Ophthalmology and Visual Science; Michael Pro, MD, Study Director — Wills Eye Institue; Steven Vold, MD, Study Director — Boozman-Hof Eye Clinic; Angelo Tanna, MD, Study Director — Northwestern Memorial Hospital; David Godfrey, MD, Study Director — Glaucoma Associates of Texas; Paul Sidoti, MD, Study Director — New York Eye and Ear Infirmiry
Locations (8):
- United States (8):
  - VoldVision-Holf Eye Clinic, Rogers, Arkansas
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Institue of Ophthalmology and Visual Science, Newark, New Jersey
  - Glaucoma Associates of New York, New York, New York
  - New York Eye and Ear Infirmary, New York, New York
  - Dean McGee Eye Institue, Oklahoma City, Oklahoma
  - Wills Eye Institue, Philadelphia, Pennsylvania
  - Glaucoma Associates of Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740
- [Derived] Tanna AP, Rademaker AW, de Moraes CG, Godfrey DG, Sarkisian SR Jr, Vold SD, Ritch R. Collagen matrix vs mitomycin-C in trabeculectomy and combined phacoemulsification and trabeculectomy: a randomized controlled trial. BMC Ophthalmol. 2016 Dec 29;16(1):217. doi: 10.1186/s12886-016-0393-z. PMID 28034308